CLINICAL TRIAL: NCT06996652
Title: An Exploratory Study of the Potential for Rational Immune System Manipulation to Prevent Emergence of Synucleinopathy Manifestations in Persons With REM Sleep Behavior Disorder (RBD)
Acronym: PRISMS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Marcus Foundation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jesse Cedarbaum, Professor of Neurology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2000038476; 2000038206 (Other: Yale); YPD-001 (Other: Yale)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Parkinson Disease Related Pattern
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Participants with REM sleep behavior disorder (RBD) who are at risk for developing motor and/or cognitive symptoms of Parkinson's disease or Lewy Body Dementia at up to 15 sites in the United States and Canada
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study sponsor and the investigational team will remain masked. An un-masked statistician and pharmacovigilance team will monitor safety of the study participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adalimumab (Experimental): Participants in this arm will receive Adalimumab every 2 weeks for up to 2 years
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Participants in this arm will receive matching placebo every 2 weeks for up to 2 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — 40 mg self-administered subcutaneously using a pre-filled syringe (PFS) every 2 weeks for up to 2 years
  Arms: Adalimumab
Drug: Placebo — 40 mg matching placebo self-administered subcutaneously using a pre-filled syringe (PFS) every 2 weeks for up to 2 years
  Arms: Placebo

SUMMARY:
This is a phase 2 study to assess the ability of adalimumab as compared to placebo to reduce or prevent progression of synuclein-related neurodegeneration in persons with idiopathic REM Sleep Behavior Disorder (RBD). The Primary Endpoint will be change from baseline in expression of the Parkinson Disease Related Pattern (PDRP) will be assessed using change in 18-flurodeoxyglucose (FDG) Positron Emission Tomography (PET) imaging.

DETAILED DESCRIPTION:
Primary Objective: To assess the ability of adalimumab as compared to placebo to reduce or prevent progression of synuclein-related neurodegeneration in persons with idiopathic REM Sleep Behavior Disorder (RBD).

Secondary Objective, Safety: Safety will be assessed by monitoring the Incidence of adverse events, clinical laboratory abnormalities, serious infections, signs and symptoms suggestive of new onset demyelinating disease, incidence of new demyelinating lesions on brain MRI scan and number of study participants who develop serum anti-adalimumab antibodies (ADAs).

Secondary Objective, Clinical: To assess the effect of adalimumab treatment on change in clinical measures presumptively related to underlying neurodegeneration. The key secondary endpoint of interest will be a composite outcome. A study participant will be considered to have met the study endpoint upon the attainment of at least 1 of the following milestones at 2 consecutive study visits at least 3 months apart:

* Increase from baseline of > 2 points on the combined MDS-UPDRS Parts 1b and 2, OR
* Increase from baseline in MDS-UPDRS Part III motor score > 4 points, OR
* Decrease from baseline in MoCA of > 3 points

Additional (or Exploratory) Objectives:

* To evaluate the pharmacodynamic effect of adalimumab on biomarkers of immune system dysfunction in RBD patients to predict response to treatment
* To evaluate the effect of adalimumab on selected biomarkers reflective of neurodegeneration
* To evaluate effects of adalimumab treatment on selected measures of quality of life

After a 12-week screening period, subjects will be randomized 1:1 to receive active or placebo treatment. Thereafter, subjects will be seen in clinic at 4, 12 and 26 weeks after their initial dose, and then at approximately 26-week intervals up to Week 96. A safety follow-up visit will occur 70 days after the last dose of study treatment. At specified visits, safety and clinical and biomarker assessments will be obtained, and study medication will be dispensed. Quantitative motor and cognitive assessments will be completed at home at intervals between in-person study visits.

At 6-monthly intervals, subjects will be given a body-worn sensor that they will wear for 7 days to record patterns of activity during sleep and wakefulness.

Subjects who meet one of the clinical secondary endpoints will remain in the study until its termination.

Approximately 25 subjects in each treatment group will be enrolled in an Cerebrospinal Fluid (CSF) biomarker sub-study. Subjects in this sub-study: Individuals participating in the CSF sub-study will undergo lumbar punctures at baseline and at yearly intervals, thereafter, to assess the effects of adalimumab on biomarkers of immune processes and neurodegeneration in the CSF.

ELIGIBILITY:
Inclusion Criteria:

* Males, or females who are either

  1. post-menopausal or otherwise not of child-bearing potential, defined as either 1) having had no menses for 12 or months without an alternative medical cause or explanation or 2) having undergone a surgical procedure (hysterectomy, bilateral tubal ligation) that prevents conception, or
  2. practicing adequate contraception. Female subjects of childbearing potential must practice at least 1 protocol-specified method of birth control, that is effective from 30 days before baseline (or earlier) through at least 150 days after the last dose of the study drug. Female subjects of non-childbearing potential do not need to use birth control.
* Diagnosis of idiopathic REM sleep behavior disorder Diagnosis of idiopathic REM Sleep Behavior Disorder (RBD) based upon:

  1. History of Dream Enactment Behavior during sleep and
  2. Evidence of REM sleep without muscle atonia based upon polysomnogram obtained in a qualified sleep laboratory, consistent with ICSD-3 Diagnostic Criteria for RBD
* Hyposmia, defined as score < 15th percentile for age-and gender-specific normal values
* Not diagnosed with motor parkinsonism or Lewy body dementia
* Have a MoCA score at screening and baseline >23
* Able to speak, read and write fluently in English, Spanish, or French
* Subject must be willing and able to attend all study visits as required by the study protocol
* Subject must have a study partner who is in regular contact with the subject and can accompany the subject to clinic visits and report on subject's functional status
* Subject must be able to self-inject study drug regularly or have a study partner who is available, willing and able to do so
* Subject must be able to understand the study requirements and provide written informed consent

Exclusion Criteria:

* Alternative explanation or etiology for the presence of RBD (e.g. narcolepsy)
* Other than RBD, neurologic or medical disorder which may impair cognition including: head trauma, seizure disorder, neurodegenerative disease, hydrocephalus, cerebral/spinal hematoma, inflammatory disease, CNS infection (e.g., encephalitis or meningitis), neoplasm, toxic exposure, metabolic disorder (including hypoxic or hypoglycemic episodes), or endocrine disorder, or any significant medical conditions that, in the opinion of the investigator, would prohibit their participation in the study.
* As assessed by the central reader, MRI evidence of (a) more than three lacunar infarcts, (b) territorial infarct or macroscopic hemorrhage, or (c) deep white matter lesions corresponding to a Fazekas score of 3
* Any contra-indication to undergo MRI, as judged by local PI or radiologist, including but not limited to presence of pacemaker, aneurysm clips, artificial heart valves, ear implants, ventriculoperitoneal shunt, foreign metal objects in the eyes, skin or body or any other circumstance which would contra-indicate an MRI scan or impair MRI image quality, or history of claustrophobia or of not tolerating MRI scanning procedures
* History or active presence of any of the following neurological, psychiatric or medical conditions:

  1. Large vessel stroke
  2. Peripheral or CNS demyelinating disease
  3. Chronic and/or recurrent fungal, bacterial or opportunistic infections
  4. Myocardial infarction or unstable angina within the previous 12 months
  5. Clinically relevant or significant ECG abnormalities, including ECG with QT interval corrected for heart rate using Fridericia's formula (QT interval corrected for heart rate using Fridericia's formula) > 450 msec (males) or > 470 msec (females).
  6. Congestive heart failure, NYHA Class 3 or 4
  7. Autoimmune disease (e.g., Systemic Lupus Erythematosis (SLE), or symptoms suggestive of a lupus-like syndrome, multiple sclerosis, rheumatoid arthritis, Type 1 diabetes mellitus, inflammatory bowel disease, psoriasis, etc.)
  8. Immunocompromised systemically due to continuing effects of immune suppressing medication
  9. Current or previous hepatitis B infection (defined as positive test for hepatitis B surface antigen (HbSAg) and/or hepatitis B core antibody (anti-HBc).

     Subjects with immunity to hepatitis B (if due to natural infection defined as negative HBsAg, positive hepatitis B antibody (anti-HBs) and positive anti-HBc; if due to vaccination defined as negative HBsAg, negative anti-HBc and positive anti-HBs are eligible to participate in the study For patients with resolved HBV infection, if anti-HBc negative, HBV DNA testing is needed prior to initiating study drug
  10. History or positive test at Screening for hepatitis C virus antibody (anti-HCV) in the absence of treatment resulting in cure
  11. History or positive test at Screening for human immunodeficiency virus (HIV)
  12. History of untreated or incompletely treated tuberculosis or a positive tuberculosis IGRA test.
  13. History of malignancy other than successfully treated, non-metastatic cutaneous squamous or basal cell carcinoma or localized carcinoma in situ of the cervix
  14. Major depressive episode requiring initiation of medication or hospitalization within the previous 90 days
  15. Seated blood pressure > 150/90 on 3 separate determinations
  16. Presence of hallucinations or delusions
  17. Psychiatric disorder (schizophrenia, schizoaffective disorder, etc.) associated with psychosis
  18. Active infection(s) requiring treatment with intravenous anti-infectives within 30 days, or oral/intramuscular anti-infectives within 14 days prior to baseline
  19. Major surgery within 12 weeks of screening
  20. Blood donation of 1 unit or more within 8 weeks prior to the first dose of study medication
* Any of the following laboratory abnormalities at Screening

  1. Screening values for hemoglobin < 12 g/d for men or < 11 g/dL for women or other clinically significant hematological abnormality
  2. Any serum chemistry value (e.g., AST, ALT, alkaline phosphatase, CK, total bilirubin etc. > 2x the upper limit of normal on 2 successive determinations less than 2 weeks apart
  3. Serum creatinine above the ULN or eGFR < 60 mL/min/1.73 m2
  4. Platelet count, INR, PT or PTT not within the normal range or other risk for increased or uncontrolled bleeding
* Any other significant medical conditions that, in the opinion of the investigator, would prohibit participation in the study, including inability to tolerate the MRI scan
* For subjects agreeing to lumbar puncture: Presence of contra-indication to lumbar puncture as judged by local PI (e.g., known X-ray or other evidence of significant lumbar spine abnormalities or history of lumbar surgery with sequalae that would interfere with or pose risks from the procedure; platelet count below 50,000 cells/mL; need for anticoagulant or antiplatelet medications other than aspirin at a dose of < 100 mg/day or clopidogrel (see item 10 (g) below))
* Taking any of the following medications:

  1. Symptomatic anti-Parkinson agents, including but not limited to levodopa-containing preparations, dopamine agonists, monoamine oxidase inhibitors, amantadine, and adenosine receptor antagonists taken any time prior to the screening visit
  2. Cognitive enhancing agents, including but not limited to acetylcholinesterase inhibitors and memantine taken any time prior to the screening visit
  3. Stimulant medications, including but not limited to lisdexamphetamine, dextroamphetamine/amphetamine (Adderall) and methylphenidate taken at any time prior to the screening visit
  4. Antipsychotic agents, including pimavanserin
  5. Antidepressant medications whose dose has not been stable for at least 90 days
  6. Use of any of the following medications within 12 months prior to Screening: Immunosuppressant medications, including chronic corticosteroids, anakinra and abatacept
  7. Any previous use of injected or infused antibody therapies, including but not limited antibodies directed against TNF, anti-IL-6, natalizumab, rituximab, conventional or targeted DMARD agents
  8. For subjects agreeing to undergo lumbar puncture: Anticoagulant or anti-platelet medications including warfarin, heparinoids and direct coagulation factor inhibitors (e.g., apixaban, dabigatran, rivaroxaban) within 90 days of the planned first dose of study drug; either aspirin at a dose of <¬ 100 mg/day or clopidogrel at a dose of 75 mg/day, but use of both in combination is permitted.
  9. Received any live vaccine, with the exception of non-replicating live viral vaccines such as Jynneos vaccine, within 30 days prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 70 days after the last dose of study drug.
* History of an allergic reaction or significant sensitivity to adalimumab or constituents of the study drug (and its excipients) and/or other products in the same class
* Participation in any other interventional clinical trial, or treatment with any investigational drug or investigational use of an approved therapy within 30 days (or 5 half-lives of such agent) prior to the first Screening visit.
* History of drug or alcohol abuse within the last 5 years (including cannabis use disorder)
* Positive urine drug test at screening
* Unwillingness or inability to comply with study requirements, including self-administration of study medication, or history of noncompliance in prior clinical trials

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in Parkinson Disease Related Pattern (PDRP) expression | Baseline and Week 96
  Change from Baseline to Week 96in the expression of the Parkinson Disease Related Pattern (PDRP) assessed by 18-flurodeoxyglucose (FDG) Positron Emission Tomography (PET).

SECONDARY OUTCOMES:
Percentage of participants that experience adverse events | up to Week 96
  Percentage of participants that experience any adverse event
Percentage of participants with clinical laboratory abnormalities | up to Week 96
  Percentage of participants with any clinical laboratory abnormalities
Percentage of participants with possible new onset of disease | up to Week 96
  Percentage of participants with serious infections and/or signs and symptoms suggestive of new onset demyelinating disease
Percentage of participants with new onset of disease | up to Week 96
  Percentage of participants with new demyelinating lesions on brain MRI scan
Percentage of participants with serum anti-adalimumab antibodies (ADAs) | up to Week 96
  Percentage of participants who develop serum anti-adalimumab antibodies (ADAs)
Number of participants that meet study endpoint | up to Week 96
  This is a composite clinical outcome. A study participant will be considered to have met the study endpoint upon the attainment of at least 1 of the following milestones at 2 consecutive study visits at least 3 months apart:
  * Increase from baseline of > 2 points on the combined MDS-UPDRS Parts 1b and 2, OR
  * Increase from baseline in MDS-UPDRS Part III motor score > 4 points, OR
  * Decrease from baseline in MoCA of > 3 points

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cedarbaum, MD, Principal Investigator — Yale University
Locations (1):
- Yale Medicine, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data not considered PHI and permitted to be released per participants' consent will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years after completion of the trial and after publication of the primary study manuscript
Access Criteria: Researchers who provide a methodologically sound proposal